CLINICAL TRIAL: NCT04966338
Title: A Phase III, Randomized, Two-armed, Double-blind, Parallel, Active-controlled Clinical Trial to Evaluate Equivalency of the Efficacy and Safety of Ocrelizumab (CinnaGen, Iran) in Comparison to Reference Product, Ocrevus® (Roche, Switzerland) in Patients With Relapsing Multiple Sclerosis
Brief Title: Efficacy and Safety of Xacrel® (Ocrelizumab) in Participants With Relapsing Remitting Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cinnagen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OCR.CIN.MS.96.III
Record Dates: First submitted 2021-06-27; First posted 2021-07-19 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Multiple Sclerosis; Relapsing-Remitting
Keywords: RRMS; Annualized Relapse Rate; Monoclonal; Humanized; Ocrelizumab
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ocrelizumab (CinnaGen, Iran) (Experimental): Ocrelizumab (CinnaGen, Iran) 600 mg (given as dual infusions of ocrelizumab 300 mg on Days 1 and 15 of the first 24-week treatment cycle and as single infusions of 600 mg on Day 1 for each 24-week treatment cycle, thereafter) every 24 weeks.
  Interventions: Biological: Ocrelizumab (CinnaGen, Iran)
- Ocrelizumab (Roche, Switzerland) (Active Comparator): Ocrelizumab (Roche, Switzerland) 600 mg (given as dual infusions of ocrelizumab 300 mg on Days 1 and 15 of the first 24-week treatment cycle and as single infusions of 600 mg on Day 1 for each 24-week treatment cycle, thereafter) every 24 weeks.
  Interventions: Biological: Ocrelizumab (Roche, Switzerland)

INTERVENTIONS:
Biological: Ocrelizumab (CinnaGen, Iran) — Ocrelizumab (CinnaGen, Iran) will be administered via intravenous (IV) infusion.
  Other Names: Xacrel®
  Arms: Ocrelizumab (CinnaGen, Iran)
Biological: Ocrelizumab (Roche, Switzerland) — Ocrelizumab (Roche, Switzerland) will be administered via intravenous (IV) infusion.
  Other Names: Ocrevus®
  Arms: Ocrelizumab (Roche, Switzerland)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Ocrelizumab produced by CinnaGen compared with Ocrevus® (Roche, Switzerland) in subjects with relapsing remitting multiple sclerosis (RRMS).

All the participants will receive one of the following regimens:

Ocrelizumab (CinnaGen) or Ocrevus® (Roche, Switzerland) ,600 mg (given as dual infusions of ocrelizumab 300 mg on Days 1 and 15 of the first 24-week treatment cycle and as single infusions of 600 mg on Day 1 for each 24-week treatment cycle, thereafter) every 24 weeks.

The primary objective of this study is to verify the equivalency of Ocrelizumab (CinnaGen) versus Ocrevus® (Roche, Switzerland) in reducing the annualized relapse rate (ARR) in participants with relapsing remitting multiple sclerosis (RRMS) at 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written, informed consent and to be compliant with the schedule of protocol assessments.
2. Ages 18-55 years at screening, inclusive.
3. Diagnosis of MS, in accordance with the revised McDonald criteria (2010).
4. At least two relapses having occurred within the past 2 years or one relapse within the past 12 months prior to screening.
5. Neurological stability for ≥ 30 days prior to both screening and baseline.
6. EDSS, at screening, from 0 to 5.5 inclusive.
7. Patients of reproductive potential must use reliable means of contraception.

Exclusion Criteria:

1. Diagnosis of primary progressive MS.
2. Disease duration of more than 10 years in patients with an EDSS ≤ 2.0 at screening.
3. Inability to complete an MRI (contraindications for MRI include but are not restricted to claustrophobia, weight ≥ 140 kg, pacemaker, cochlear implants, presence of foreign substances in the eye, intracranial vascular clips, surgery within 6 weeks of entry into the study, coronary stent implanted within 8 weeks prior to the time of the intended MRI, etc).
4. Known presence of other neurological disorders which may mimic MS including but not limited to: neuromeylitis optica, Lyme disease, untreated vitamin B12 deficiency, neurosarcoidosis and cerebrovascular disorders.
5. Pregnancy or lactation.
6. Any concomitant disease that may require chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study.
7. History or currently active primary or secondary immunodeficiency.
8. Lack of peripheral venous access.
9. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies.
10. Significant or uncontrolled somatic disease or any other significant disease that may preclude patient from participating in the study such as Congestive heart failure (NYHA III or IV functional severity).
11. Known active bacterial, viral, fungal, mycobacterial infection or other infection, excluding fungal infection of nail beds.
12. Infection requiring hospitalization or treatment with I.V. antibiotics within 4 weeks prior to baseline visit or oral antibiotics within 2 weeks prior to baseline visit.
13. History or known presence of recurrent or chronic infection (e.g., hepatitis B or C, HIV).
14. History of progressive multifocal leukoencephalopathy (PML)
15. History of malignancy, including solid tumors and hematological malignancies, except basal cell carcinoma, in situ squamous cell carcinoma of the skin, and in situ carcinoma of the cervix of the uterus that have been previously completely excised with documented, clear margins.
16. History of alcohol or drug abuse within 24 weeks prior to baseline.
17. History or laboratory evidence of coagulation disorders.
18. Receipt of a live vaccine (BCG, MMR, VZV, polio, yellow fever and some influenza vaccine) within 6 weeks prior to baseline. In rare cases when patient requires vaccination with a live vaccine, the screening period may be extended but cannot exceed 8 weeks.
19. Treatment with any investigational agent within 24 weeks of screening (Visit 1) or five half-lives of the investigational drug (whichever is longer).
20. Contraindications to or intolerance of oral or i.v. corticosteroids, including methylprednisolone administered i.v.
21. Treatment with dalfampridine unless on stable dose for ≥ 30 days prior to screening. Patients should remain on stable doses throughout the 48 weeks' treatment period.
22. Previous treatment with B-cell targeted therapies (i.e. rituximab, ocrelizumab, atacicept, belimumab or ofatumumab).
23. Systemic corticosteroid therapy within 4 weeks prior to screening.
24. Any previous treatment with anti-CD4, cladribine, mitoxantrone, daclizumab, teriflunomide, laquinimod, total body irradiation or bone marrow transplantation.
25. Treatment with cyclophosphamide, azathioprine, mycophenolate mofetil (MMF), cyclosporine, methotrexate or natalizumab within 24 months prior to screening. Patients previously treated with natalizumab will be eligible for this study only if duration of treatment with natalizumab was < 1 year.
26. Treatment with fingolimod or dimethyl fumarate (DMF) within 4 weeks prior to screening. Only patients with T lymphocyte count ≥ LLN will be eligible for this study.
27. Treatment with I.V. immunoglobulin within 12 weeks prior to baseline.
28. Positive serum β hCG measured at screening.
29. Positive screening tests for hepatitis B
30. CD4 count < 300/μL.
31. AST/SGOT or ALT/SGPT ≥ 2.0 Upper Limit of Normal (ULN).
32. Platelet count <100,000/μL (<100 x 109/L).
33. Levels of serum IgG 18% below the LLN.
34. Levels of serum IgM 8% below the LLN.
35. Total neutrophil count <1.5 x 10^3/μL.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Annualized Relapse Rate at 48 weeks | 48 weeks
  Total number of confirmed relapses divided by the total number of days on study A relapse is defined as the appearance of a new or worsening of a previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding relapse. The abnormality must be present for at least 24 hours and occur in the absence of fever or infection

SECONDARY OUTCOMES:
Time to onset of sustained disability progression for at least 12 weeks | Baseline up to Week 96
  Disability progression is defined as an increase in the Expanded Disability Status Scale (EDSS) score of:
  A) At least a 1.5-point increase in patients with a baseline score of 0 B) At least a 1.0-point increase on the EDSS in patients with a baseline score of 0<EDSS≤5.5 C) At least a 0.5-point increase on the EDSS in patients with a baseline score of >5.5
  The EDSS scale ranges from 0 (normal neurological exam) to 10 (death due to multiple sclerosis)
Time to onset of sustained disability progression for at least 24 weeks | Baseline up to Week 96
  Disability progression is defined as an increase in the Expanded Disability Status Scale (EDSS) score of:
  A) At least a 1.5-point increase in patients with a baseline score of 0 B) At least a 1.0-point increase on the EDSS in patients with a baseline score of 0<EDSS≤5.5 C) At least a 0.5-point increase on the EDSS in patients with a baseline score of >5.5
  The EDSS scale ranges from 0 (normal neurological exam) to 10 (death due to multiple sclerosis)
Proportion of relapse-free patients by 96 weeks | Week 96
  A relapse is defined as the appearance of a new or worsening of a previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding relapse. The abnormality must be present for at least 24 hours and occur in the absence of fever or infection
Total number of new Gadolinium (Gd)-enhancing lesions as detected by brain MRI | Baseline up to Week 96
  Sum of the individual number of (Gd)-enhancing lesions at Weeks 24, 48, and 96
Total number of new, and/or enlarging T2 hyperintense lesions as detected by brain MRI | Baseline up to Week 96
  Sum of the individual number of new, and/or enlarging T2 hyperintense lesions at Weeks 24, 48, and 96
Change in total T2 lesion volume as detected by brain MRI from baseline to week 96 | Baseline up to Week 96
Number of Participants With Adverse Events (AEs) | Baseline up to Week 96
  Intensity, seriousness and causality assessment of observed AEs, and abnormal laboratory findings every 12 weeks.
Number of Participants With Infusion Related Reactions (IRRs) | Baseline up to Week 96
  Assessment of IRRs every 24 weeks
Immunogenicity Assessment | Baseline up to Week 96
  Number of participants positive for anti-drug antibodies at weeks 24, 48 and 96

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Ali Sahraian, professor, Principal Investigator — Neurologist/MS Research Center, Neuroscience Institute ,Tehran University of Medical Sciences
Locations (15):
- Iran (15):
  - Qaem International Hospital, Rasht, Gilan Province
  - Qaem Hospital, Mashhad, Khorasan Razavi
  - Golestan Hospital, Ahvāz, Khozestan
  - Bouali Hospital, MS Clinic, Sari, Mazandaran
  - Sina Hospital, Hamadan
  - Ayatollah Kashani Hospital, MS Clinic, Isfahan
  - Shafa Hospital, Kerman
  - Imam Reza Hospital, Kermanshah
  - Dr. Nikseresht's office, Shiraz
  - Namazi Hospital, Shiraz
  - Imam Reza Hospital Department of Neurology, Tabriz
  - Amir Alam Hospital, Tehran
  - Imam Hossein Hospital, MS Clinic, Tehran
  - Imam Khomeini Hospital, Tehran
  - Sina Hospital, MS Research Center, Tehran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sahraian MA, Abolfazli R, Shaygannejad V, Ashtari F, Majdinasab N, Navardi S, Baghbanian SM, Sedighi B, Naser Moghadasi A, Nahayati MA, Ghalyanchi Langroodi H, Mohammadianinejad SE, Beladi Moghadam N, Ayromlou H, Nikseresht A, Ghiasian M, Razazian N, Asadollahzadeh E, Sabzvari A, Kafi H, Albooyeh S. Evaluating efficacy and safety of ocrelizumab biosimilar (Xacrel) compared to the originator (Ocrevus) in relapsing multiple sclerosis: a phase III, randomized, equivalency, clinical trial. Sci Rep. 2024 Oct 22;14(1):24921. doi: 10.1038/s41598-024-75745-y. PMID 39438591